CLINICAL TRIAL: NCT00852436
Title: Efficacy of Pregabalin in the Treatment of Orofacial Neuropathic Pain
Brief Title: Pregabalin and Orofacial Neuropathic Pain
Acronym: Pregabalin-Dao
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty to recruit patients
Sponsor: University of Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Thuan Dao, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dao-Watson Pregabalin
Record Dates: First submitted 2008-11-06; First posted 2009-02-27 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2010-11

CONDITIONS: Neuropathic Pain; Orofacial Pain
Keywords: neuropathic pain; orofacial pain; clinical trials; pregabalin; randomized controlled trial
MeSH Terms: conditions — Neuralgia; Facial Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pregabalin capsules in 75 mg, administered orally one (or two, or four) capsule(s), twice daily. Dosing increment from 150, 300, to 600mg/day at weekly intervals.
  Interventions: Drug: pregabalin
- 2 (Placebo Comparator): Placebo capsules in 75 mg, administered orally one (or two, or four) capsule(s), twice daily. Dosing increment from 150, 300, to 600mg/day at weekly intervals.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — Pregabalin capsules in 75 mg,dosing increment from 150, 300, to 600mg/day at weekly intervals,administered orally one (or two, or four) capsule(s), twice daily. Fixed schedule of dosing increment from 150, 300, to 600mg/day at weekly intervals, until the highest tolerated dose has been reached. A single downward dose titration will be allowed depending on tolerability, after which the patient will remain on this dosage for the rest of the study.
  Other Names: Lyrica
  Arms: 1
Drug: placebo — Placebo capsules in 75 mg,dosing increment from 150, 300, to 600mg/day at weekly intervals,administered orally one (or two, or four) capsule(s), twice daily. Fixed schedule of dosing increment from 150, 300, to 600mg/day at weekly intervals, until the highest tolerated dose has been reached. A single downward dose titration will be allowed depending on tolerability, after which the patient will remain on this dosage for the rest of the study.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether pregabalin can decrease pain and improve quality of life in patients who have nerve pain on the mouth or the face

DETAILED DESCRIPTION:
Neuropathic pain (NP) is defined as pain initiated or caused by a primary lesion or dysfunction in the nervous system. At the trigeminal area where somatosensory nerves are often damaged during dental /maxillofacial interventions, post-operative orofacial neuropathic pain (OFNP) estimated treated prevalence/incidence rates were ~3-12%, with 83% of patients reporting that OFNP started with a dental treatment. Although OFNP is a burden for the society, and a major cause of chronic distress, disability and expenditure of medical resources, clinical trials that assess efficacy of its treatment are scarce. Until today, treatments of OFNP are extrapolated from those issued for neuropathic pain in other body sites. This clinical trial will be the first to evaluate the efficacy, safety, and tolerance of pregabalin in the treatment of OFNP. Based on the results obtained for neuropathic pain on non trigeminal areas, we expect to see positive results, and to provide evidence for effective management of OFNP with an anticonvulsant such as pregabalin.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older, males and females
* history of dental and/or maxillofacial treatment/surgery that may cause nerve injury (e.g. root canal treatment, implant placement, deep restorations, tooth extractions, injection of anesthetics)
* patients who score 12 on the validated self-report version of the Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS; Bennett et al. 2005) for extra-oral sites, or 9 for intra-oral sites (the scoring for extra-oral sites is taken as suggested; for intra-oral sites, the 5-point scoring for question 2 has been removed and the score proportionally adjusted, since it is difficult for patients to see color changes in their mouth)
* pain rated 4 or more on a numerical scale (0 being no pain, 10 being the most intense pain imaginable), on a daily basis
* pain lasting more than 6 months
* absence of identifiable organic lesion, inflammation or infection
* normal serum creatinine
* reports that current and previous pain medications failed to provide adequate relief (e.g., analgesic, non-steroidal anti-inflammatories, opioids, antidepressants)
* if currently using medication, acceptance of a wash-out period of at least one week, during which only Tylenol can be used as rescue medication
* able to use the Palm handheld device to report daily pain

Exclusion Criteria:

* lactating, pregnancy (potentially child bearing patients need to have a referral from family physician stating that the patient is not expecting or to be using contraception)
* renal impairment or renal failure (contra-indication to pregabalin)
* congestive heart failure or liver disease
* currently suffering from trigeminal neuralgia
* history of mental disorder, widespread pain or other severe pain conditions that may confound the pain assessment (e.g. depression, chronic fatigue, migraine headaches, fibromyalgia, severe chronic pain conditions)
* intolerance or allergy to gabapentin and pregabalin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 12 weeks

SECONDARY OUTCOMES:
Pain unpleasantness | 12 weeks
Quality of life using the modified short form of Oral health Impact Profile | 12 weeks
Anxiety and Depression measured with the Hospital Anxiety and Depression Rating scae | 12 weeks
Patient global impression of change | 12 weeks
Proportion of patients with 30% and 50% reduction of pain | 2 years
Side effects | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thuan Dao, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Dr. P. Watson's office, Etobicoke, Ontario
  - University of Toronto, Toronto, Ontario